CLINICAL TRIAL: NCT02888171
Title: Impact of Ferric Citrate vs Ferrous Sulfate on Iron Parameters and Hemoglobin in Individuals With Moderate to Severe Chronic Kidney Disease (CKD) With Iron Deficiency
Brief Title: Impact of Ferric Citrate vs Ferrous Sulfate on Iron Parameters and Hemoglobin in Individuals With CKD and Iron Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Orlando M. Gutierrez, MD, MMSc, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F160318006
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Chronic Kidney Disease; Iron Deficiency; Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Iron Deficiencies; Anemia | interventions — ferric citrate; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ferric citrate (Experimental): Participants randomized to the ferric citrate arm will receive 2 grams of ferric citrate three times a day with each meal.
  Interventions: Drug: ferric citrate
- ferrous sulfate (Active Comparator): Participants randomized to the ferrous sulfate arm will receive 325 mg of ferrous sulfate three times a day
  Interventions: Drug: ferrous sulfate

INTERVENTIONS:
Drug: ferric citrate — Participants randomized to the ferric citrate arm will take 2 grams of ferric citrate three times a day with meals.
  Other Names: Auryxia
  Arms: ferric citrate
Drug: ferrous sulfate — Participants randomized to the ferrous sulfate arm will take 325 mg of ferrous sulfate three times a day.
  Arms: ferrous sulfate

SUMMARY:
The main objective of the study is to compare the impact of oral ferric citrate compared to standard of care oral ferrous sulfate on serum iron, percent transferrin saturation, ferritin, hepcidin and hemoglobin levels in individuals with moderate to severe chronic kidney disease (CKD) and absolute iron deficiency.

DETAILED DESCRIPTION:
Ferric citrate is an FDA-approved oral phosphorus binder that has been shown to be effective in reducing serum phosphorus and fibroblast growth factor 23 (FGF23) concentrations and increasing iron stores and hemoglobin in individuals with non-dialysis-dependent CKD who have iron-deficiency anemia. This may prove to be advantageous in individuals with pre-dialysis CKD who require iron supplementation for iron-deficiency anemia. This is because ferric citrate may not only restore iron stores in individuals who are iron deficient, but by lowering FGF23 concentrations, ferric citrate may increase local and systemic concentrations of 1,25-dihydroxyvitamin D, a powerful inhibitor of hepcidin synthesis, potentially attenuating the increase in hepcidin following oral iron supplementation. When compared to standard iron supplementation therapies (e.g., oral ferrous sulfate) that powerfully stimulate hepcidin secretion, this may then allow for greater iron bioavailability by increasing iron absorption in the gut while also reducing the degree of iron sequestration in reticuloendothelial system stores. However, little is known about the comparative effectiveness of treatment with oral ferric citrate vs. oral ferrous sulfate (currently the standard of care) in increasing iron stores and hemoglobin in iron-deficient CKD patients. If ferric citrate is shown to not only improve overall iron status, but also partially mitigate the long-term effects of iron supplementation on hepcidin secretion by increasing endogenously produced 1,25-dihydroxyvitamin D, this may indicate that ferric citrate can provide superior short- and long-term effects on iron-restricted erythropoiesis in CKD as compared to the current standard of care. The main objectives of the study are to compare the impact of ferric citrate compared to standard of care ferrous sulfate on serum iron, percent transferrin saturation (TSAT), ferritin, hemoglobin and hepcidin concentrations in individuals with moderate to severe CKD and absolute iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Moderate to severe CKD not requiring dialysis (eGFR 15 - 45 ml/min/1.73 m2 by CKD-EPI)
* Absolute iron deficiency (serum ferritin <300ng/ml and Transferrin Saturation < 30%)

Exclusion Criteria:

* Hemoglobin concentrations > 13 g/dL
* Known disorder of iron homeostasis (e.g., hemochromatosis)
* Known gastrointestinal disorder (irritable bowel disease, inflammatory bowel disease)
* Known liver disease (ALT/AST or bilirubin > 3x normal)
* Serum phosphorus concentrations < 3.0 mg/dL
* Any known cause of anemia other than iron deficiency or CKD (e.g., sickle cell anemia)
* Symptomatic gastrointestinal bleeding within 12 weeks prior to the screening visit.
* Subjects receiving any form of renal replacement therapy including hemodialysis, peritoneal dialysis, or renal transplant.
* Pregnancy or lactation in female participants
* Severe anemia defined as a hemoglobin < 8.0 g/dL for males or a hemoglobin <7.0 g/dL for females.
* Receipt of erythropoiesis stimulating agents within 4 weeks of screening.
* Receipt of intravenous iron therapy within 8 weeks of screening.
* Blood transfusion within 4 weeks of screening
* Known allergies or severe adverse reactions to previous oral iron therapy
* Current use of oral phosphorus binders.
* Current use of an active vitamin D analog

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orlando M Gutierrez, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Womack R, Berru F, Panwar B, Gutierrez OM. Effect of Ferric Citrate versus Ferrous Sulfate on Iron and Phosphate Parameters in Patients with Iron Deficiency and CKD: A Randomized Trial. Clin J Am Soc Nephrol. 2020 Sep 7;15(9):1251-1258. doi: 10.2215/CJN.15291219. Epub 2020 Jul 21. PMID 32694162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the nephrology outpatient clinics at the University of Alabama at Birmingham (UAB) from September 2016 to October 2018.
Pre-assignment Details: Participants who were taking oral iron supplements at the time of the screening visit were allowed to participate but had to undergo a wash-out period of at least 4 weeks prior to randomization.
Period: Overall Study
Arm/Group | Ferric Citrate | Ferrous Sulfate
Started | 30 | 30
Completed | 25 | 26
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Citrate | Ferrous Sulfate | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12) | 63 (11) | 62 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 17 | 33
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
body mass index [Mean (Standard Deviation); unit: kg/m^2] | 37 (8) | 36 (9) | 36 (8)
systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 136 (21) | 134 (20) | 135 (20)
diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 74 (11) | 73 (10) | 73 (10)
phosphorus [Mean (Standard Deviation); unit: mg/dL] | 3.7 (0.5) | 3.9 (0.8) | 3.8 (0.7)
calcium [Mean (Standard Deviation); unit: mg/dL] | 9.3 (0.4) | 9.3 (0.7) | 9.3 (0.6)
estimated glomerular filtration rate [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 33 (12) | 26 (14) | 31 (13)
transferrin saturation [Mean (Standard Deviation); unit: %] | 18 (6) | 19 (6) | 18 (6)
ferritin [Mean (Standard Deviation); unit: ng/ml] | 90 (70) | 100 (59) | 95 (65)
hemoglobin [Mean (Standard Deviation); unit: g/dL] | 11.4 (1) | 11.0 (1) | 11.2 (1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Ferritin From Baseline to End of Treatment
Description: The change in serum ferritin concentrations from the baseline of the study to the 12 week time point.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Ferric Citrate | Ferrous Sulfate
Number analyzed (Participants) | 28 | 29
percentage of change from baseline | 60 (17) | 30 (10)

2. Primary Outcome: Change in Transferrin Saturation From Baseline to End of Treatment
Description: The change in serum transferrin saturation from the baseline to the end of treatment
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Ferric Citrate | Ferrous Sulfate
Number analyzed (Participants) | 28 | 29
percentage of change from baseline | 40 (17) | 2 (7)

3. Secondary Outcome: Change in Hemoglobin From Baseline to End of Treatment
Description: The change in hemoglobin concentrations from the baseline visit to the 12-week time point.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Ferric Citrate | Ferrous Sulfate
Number analyzed (Participants) | 28 | 29
percentage of change from baseline | 4 (0.1) | 0 (0.1)

4. Secondary Outcome: Change in Hepcidin From Baseline to the End of Treatment
Description: The change in hepcidin concentrations from the baseline visit to the 12-week time point.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Ferric Citrate | Ferrous Sulfate
Number analyzed (Participants) | 20 | 20
percentage of change from baseline | 98 (20) | 28 (11)

5. Secondary Outcome: Change in Fibroblast Growth Factor 23 From Baseline to the End of Treatment
Description: The change in fibroblast growth factor 23 concentrations from the baseline visit to the 12-week time point.
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Ferric Citrate | Ferrous Sulfate
Number analyzed (Participants) | 28 | 29
pg/ml | -37 [-74 to 1] | -8 [-32 to 16]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Ferric Citrate | Ferrous Sulfate
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 26/30 | 24/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Citrate (N=30) | Ferrous Sulfate (N=30)
Change in stool color (Gastrointestinal disorders) | 16 (16) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 5 (5)
Constipation (Gastrointestinal disorders) | 9 (9) | 11 (11)
Anorexia (Gastrointestinal disorders) | 2 (2) | 8 (8)
Weight Loss (General disorders) | 3 (3) | 7 (7)
Weight gain (General disorders) | 5 (5) | 8 (8)
Fatigue (General disorders) | 6 (6) | 3 (3)
Infection (Infections and infestations) | 5 (5) | 1 (1)
Eye pain (Eye disorders) | 2 (2) | 5 (5)
Vision changes (Eye disorders) | 4 (4) | 4 (4)
Nasal congestion (Ear and labyrinth disorders) | 3 (3) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 5 (5)
GERD (Gastrointestinal disorders) | 3 (3) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
edema (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Headache (General disorders) | 2 (2) | 6 (6)
change in smell (Ear and labyrinth disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT02888171/Prot_SAP_000.pdf